

Comparing the Effect of Early Childhood Caries Treatment Procedures Under General and Local anesthesia on the Quality of Life of Young Children

Statistical Analysis plan March 2021

## Statistical Analyses

The data were subjected to bivariate and multivariable analysis. Between both groups, the mean and standard deviation (SD) values of age and dft index were computed. For all categorical variables, the frequencies and percentages were calculated. The Chi-square test of significance was used to assess the difference in proportion of study participants in the LA and DGA groups with regards to each of the assessed variable. Because the data was not distributed normally, the subsequent tests of associations were performed using non-parametric tests. A Friedman test was carried out to examine the mean difference between the LA and DGA groups at the baseline, one-week and one-month timelines. All tests were set at 5% significance and the analyses were performed using SPSS version 24 (IBM, USA). Intention-to-treat principle was observed, and all randomized participants were analyzed according to the group that they were originally allocated.